CLINICAL TRIAL: NCT01544803
Title: Randomized Controlled Trial of eScreen for Problematic Alcohol Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/308-31/5A
Record Dates: First submitted 2011-10-27; First posted 2012-03-06 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Problematic AOD Use
Keywords: Randomized Controlled Trial; Alcohol; Internet; Screening; Brief intervention; Personalized feedback

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention)
- Web based self-monitoring (Experimental)
  Interventions: Behavioral: eScreen
- Web based self-help (Active Comparator)
  Interventions: Behavioral: Alkoholhjalpen

INTERVENTIONS:
Behavioral: eScreen — The eScreen brief Internet intervention for problematic alcohol and drug use offers self-screening, in-depth self-reporting, personalized feedback and treatment recommendations as well as an electronic diary. Progress over time is shown in diagrams detailing consumption levels.
  Other Names: www.escreen.se
  Arms: Web based self-monitoring
Behavioral: Alkoholhjalpen — An extensive Internet intervention for problematic alcohol use, Alkoholhjalpen,provides CBT- and MI-based psycho-education with a solution-oriented focus, electronic diary and moderated chat-forum.
  Other Names: www.alkoholhjalpen.se
  Arms: Web based self-help

SUMMARY:
Objectives: This study compares the efficacy of eScreen and Alkoholhjalpen in a three-armed randomized controlled design, measuring outcomes in terms of changes in problematic alcohol use up to one year after study recruitment. The eScreen brief Internet intervention for problematic alcohol and drug use offers self-screening, in-depth self-reporting, personalized feedback and treatment recommendations as well as an electronic diary. Progress over time is shown in diagrams detailing consumption levels. A more extensive Internet intervention for problematic alcohol use, Alkoholhjalpen,provides CBT- and MI-based psycho-education with a solution-oriented focus, electronic diary and moderated chat-forum.

Method: Participants with problematic alcohol use (AUDIT >7 for men and >5 for women) are randomized into one of three groups: T1, eScreen referral (n=211); T2, Alkoholhjalpen referral (n=211); Control group (n=211). Outcomes on alcohol use as well as health-related symptoms are assessed after 3, 6 and 12 months.

The first hypothesis is that all three groups will reduce their alcohol consumption and alcohol-related problems at follow-ups compared to the baseline level. The second hypothesis is that there will be no differences between participants in the eScreen and the Alkoholhjalpen group in reduction of alcohol consumption and alcohol-related problems at follow-ups. The third hypothesis is that participants in the eScreen and the Alkoholhjalpen group will show a greater reduction in alcohol consumption and alcohol-related problems compared to the control group (no intervention) at follow-ups. For a greater understanding of the study results possible other interventions received by the study participants for their problematic alcohol use during these 12 months of study participation will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Problematic alcohol use. AUDIT>7 for men and AUDIT>5 for women

Exclusion Criteria:

* Drug use DUDIT>0
* Unproblematic alcohol use, AUDIT<8 for men and AUDIT<6 for women

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in the total AUDIT-C score | 3, 6 and 12 months
  The primary outcome measure for this trial was the change in the total AUDIT score for the first three AUDIT questions, as a measure of alcohol consumption only, referred to as the AUDIT-C.

SECONDARY OUTCOMES:
AUDIT | 3, 6 and 12 months
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems).

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Clinical Neuroscience, Stockholm, Sweden

REFERENCES:
- [Background] Sinadinovic K, Berman AH, Hasson D, Wennberg P. Internet-based assessment and self-monitoring of problematic alcohol and drug use. Addict Behav. 2010 May;35(5):464-70. doi: 10.1016/j.addbeh.2009.12.021. Epub 2010 Jan 4. PMID 20092953
- [Background] Sinadinovic K, Wennberg P, Berman AH. Population screening of risky alcohol and drug use via Internet and Interactive Voice Response (IVR): a feasibility and psychometric study in a random sample. Drug Alcohol Depend. 2011 Mar 1;114(1):55-60. doi: 10.1016/j.drugalcdep.2010.09.004. Epub 2010 Oct 27. PMID 21030164
- See also: For research group profile search Berman — http://ki.se/
- See also: Web based self-monitoring site — http://www.escreen.se
- See also: Web based self-help site — http://www.alkoholhjalpen.se